CLINICAL TRIAL: NCT00848328
Title: A Phase II Trial of the Combination of Lenalidomide and Rituximab in Patients With Relapsed/Refractory Follicular NHL (RV 0163)
Brief Title: Lenalidomide and Rituximab in Treating Patients With Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University of California, Davis (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Joseph Tuscano, Professor, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 220942; CDR0000634775 (Other: UC Davis IRB); CELGENE-RV-PI-NHL-0163 (Other Grant/Funding Number: Celgene); UCD-197 (Other: University of California Davis)
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma
Keywords: recurrent small lymphocytic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide and Rituximab (Experimental): Rituximab 375 mg/m2/wk x 4 weeks, to begin Cycle 1, Day 15. Lenalidomide 20 mg daily, days 1-21 of a 28 day cycle, to begin Day 1 of cycle 1 and continue until disease progression.
  Interventions: Biological: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Biological: Rituximab — Injection for Intravenous Use, 375 mg/m2/wk x 4 weeks, to begin Cycle 1, Day 15.
  Other Names: Rituxan, MabThera
Drug: Lenalidomide — Supplied as 5mg capsules; Dosage: 20 mg daily, days 1-21 of a 28 day cycle, to begin Day 1 of cycle 1 and continue until disease progression.
  Other Names: REVLIMID

SUMMARY:
RATIONALE: Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving lenalidomide together with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving lenalidomide together with rituximab works in treating patients with follicular or small lymphocytic non-Hodgkin lymphoma that has relapsed or not responded to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the response rate in patients with relapsed or refractory follicular or small lymphocytic non-Hodgkin lymphoma treated with lenalidomide and rituximab.

Secondary

* To determine the time to disease progression, duration of response, and overall survival of these patients.
* To determine the tolerability of this regimen in these patients.
* To assess changes in serum cytokines before and after treatment and correlate these changes with response.

OUTLINE: This is a multicenter study.

Patients receive oral lenalidomide once daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV on days 15 and 22 of course 1 and on days 1 and 8 of course 2. Patients who do not achieve complete response after 2 courses of rituximab may receive up to 4 additional doses of rituximab once weekly for 4 weeks.

Blood samples are collected at baseline and after treatment for cytokine analysis.

After completion of study treatment, patients are followed at 30 days and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically* confirmed non-Hodgkin lymphoma, including one of the following subtypes:

  * Grade 1, 2, or 3a (> 15 centroblasts per high-power field with centrocytes present) follicular lymphoma according to WHO criteria
  * Small lymphocytic lymphoma
* NOTE: *Bone marrow biopsies as the sole means of diagnosis are not acceptable, but they may be submitted in conjunction with nodal biopsies or extra-nodal biopsies; fine-needle aspirates are not acceptable for diagnosis.
* At least one measurable lesion according to RECIST criteria

  * Measurable lymphadenopathy to follow with serial exam and/or imaging
* Relapsed or refractory disease

  * Must have evidence of disease progression during or after last treatment

    * If previously treated with rituximab, must have disease progression within 6 months of last therapy OR if there was a prior response to rituximab, rituximab must not have been given within the past 6 months
* No evidence of CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 75,000/mm³
* Serum creatinine ≤ 2.0 mg/dL
* Total bilirubin ≤ 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double method contraception for ≥ 28 days before, during, and for ≥ 28 days after completion of study therapy
* HIV negative
* Able to swallow lenalidomide
* Able to take aspirin (81 or 325 mg) daily or low molecular weight heparin as prophylactic anticoagulation
* No neuropathy ≥ grade 2
* No known active hepatitis A, B, or C
* No other malignancies within the past 5 years except treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast
* No serious medical condition, laboratory abnormality, or psychiatric illness that would preclude the patient from signing the informed consent form
* No condition, including the presence of laboratory abnormalities, that would preclude study participation or confound the ability to interpret study data
* No known hypersensitivity to thalidomide or rituximab
* No development of erythema nodosum, if characterized by a desquamating rash while taking thalidomide or similar drugs

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior anticancer therapy, including radiotherapy, hormonal therapy, or surgery
* More than 28 days since prior experimental drug or therapy
* No prior lenalidomide
* No other concurrent anticancer agents or treatments, including radiotherapy or thalidomide
* No other concurrent investigational agents
* No concurrent sargramostim (GM-CSF)
* No other concurrent antilymphoma therapy, including steroids (except for the treatment of hypersensitivity reactions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-08-25 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Response, as defined by complete response (CR), near CR, partial response, or stable disease at 4 months | 4 months
  Responses will be assessed by the Revised Working Group Response Criteria for Malignant Lymphoma. A complete response is the complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. A partial response is regression of measurable disease and no new sites of disease. Stable disease is failure to attain a complete response/partial response or progressive disease.

SECONDARY OUTCOMES:
Time to disease progression | Up to two years
  Time to progression will be measured as the time from when the patient started treatment to the time the patient is first recorded as having disease progression, or the date of death if the patient dies due to causes other than disease progression
Tolerability (type, frequency, severity, and relationship of adverse events to study treatment as assessed by NCI CTCAE v3.0) | Up to two years
Duration of response | Up to two years
  The duration of response is measured from the time measurement criteria are met for complete response/partial response(whichever status is recorded first) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
  The duration of response is measured from the time measurement criteria are first met for complete response until the first date that recurrent disease is objectively documented.
Overall survival | Up to two years
  Overall survival wil be measured as the time from start of treatment to the date of death or the last date the patient was known to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M. Tuscano, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States